CLINICAL TRIAL: NCT01776047
Title: A Randomized, Open Label, Single Dose, 2-Way Cross-over Clinical Trial to Compare the Safety and Pharmacokinetic Characteristics of Exforge® and G-0081 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G-0081_BA_I
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Male Volunteer
MeSH Terms: interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exforge® 10/160 (Amlodipine besylate 10mg / Valsartan 160mg) (Active Comparator): Exforge® 10/160
  Interventions: Drug: Exforge®
- G-0081 (Amlodipine orotate 10mg / Valsratan 160mg) (Experimental): G-0081
  Interventions: Drug: G-0081

INTERVENTIONS:
Drug: Exforge®
  Arms: Exforge® 10/160 (Amlodipine besylate 10mg / Valsartan 160mg)
Drug: G-0081
  Arms: G-0081 (Amlodipine orotate 10mg / Valsratan 160mg)

SUMMARY:
Study Design : randomized, open label, single-dose, 2-way cross-over design

Phase : Phase I

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers between the ages of 20 to 50 years old within the range of ±20% of IBW(Ideal Body Weight)
* having neither congenital/chronic diseases nor pathological symptoms/findings as results of medical examination
* doctor determines to be suitable as subjects within 4 weeks ago before administration

Exclusion Criteria:

* Hypersensitivity(or history of hypersensitivity) to amlodipine and valsartan
* Active Liver Diseases or exceed 1.5 times the normal range of AST, ALT
* Gastrointestinal diseases or surgeries that affect absorption of drug
* Excessive drinking(exceed 30g/week) and excessive caffeine(exceed 250mg/day)
* Smoking over 10 cigarettes per day

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
AUClast, Cmax | Blood gathering point : 0h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h, 96h, 144h, 192h

SECONDARY OUTCOMES:
AUCinf, Tmax, t1/2, % AUCextra | Blood gathering point : 0h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h, 96h, 144h, 192h
  AUCinf = AUClast + Clast/λz
  %AUCextra = [ (AUCinf - AUClast) / AUCinf ] ×100
  t1/2 = 0.693/λz

CONTACTS AND LOCATIONS:
Overall Officials: K S Park, MD, PhD, Principal Investigator — Head of Clinical Development, Clinical Trials Center Severance Hospital